CLINICAL TRIAL: NCT06279897
Title: Skin Rewarming After Exercise Cold Stress and Tolerance to Simulated Blood Loss
Brief Title: LBNP Tolerance With Skin Warming After Exercise Cold Stress
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, James Pearson, Associate Professor, University of Colorado, Colorado Springs
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-068
Record Dates: First submitted 2024-02-07; First posted 2024-02-28 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure; Blood Loss
Keywords: Arterial Blood Pressure; Permissive Hypotension; Cold Stress; Skin Warming; Blood Loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants will complete trial 1 at the beginning of the study. Participants will then complete trials 2 through 5 in a random, counterbalanced order.
Masking Description: Participants are blinded to the skin temperature control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin Temperature Control During Simulated Blood Loss After Exercise Cold Stress (Experimental): After exercise in the cold and participants skin will remain cold (~82°F), be returned to normal (~90°F), be slightly warmed (~93°F) or heated (~95°F) sixty seconds after the onset of LBNP.
  Interventions: Other: Skin Surface Rewarming; Other: Skin Surface Warming; Other: Skin Surface Heating; Other: Skin Surface Cooling

INTERVENTIONS:
Other: Skin Surface Rewarming — Sixty seconds after the onset of lower body negative pressure (LBNP) skin temperature will be increased to ~90°F and held here for the duration of the LBNP test.
  Other Names: Normothermic Trial
Other: Skin Surface Warming — Sixty seconds after the onset of lower body negative pressure (LBNP) skin temperature will be increased to ~93°F and held here for the duration of the LBNP test.
  Other Names: Warm Trial
Other: Skin Surface Heating — Sixty seconds after the onset of lower body negative pressure (LBNP) skin temperature will be increased to ~95°F and held here for the duration of the LBNP test.
  Other Names: Hot Trial
Other: Skin Surface Cooling — Sixty seconds after the onset of lower body negative pressure (LBNP) skin temperature will remain lowered to ~82°F for the duration of the LBNP test.
  Other Names: Cold Trial; Control Trial

SUMMARY:
Assess the effect of skin rewarming during lower body negative pressure upon arterial blood pressure and tolerance to simulated blood loss after exercise in the cold.

DETAILED DESCRIPTION:
Individuals who have experienced a hemorrhagic insult are often wrapped in a warm blanket. In individuals who have exercise in a cold environment, it is unknown how this skin warming influence tolerance to simulated blood loss and whether there is an optimal temperature to warm the skin up to in order to lower blood pressure (permissive hypotension).

After an initial study visit to examine exercise capacity (Visit 1), participants will complete four trials (Visits 2 through 5) After exercise in a cold environment, participants will have cold skin temperatures (~82°F; Visit 2). Researchers will examine how increasing skin temperature to normal (~90°F; Visit 3), warm (93°F; Visit 4) and hot (95°F; Visit 5) influences arterial blood pressure and tolerance to simulated blood loss compared to when the skin remains cold.

This project will test the hypothesis that skin rewarming to ~95°F lowers arterial blood pressure without impairing tolerance to simulated blood loss (lower body negative pressure; LBNP) relative to when the skin is kept cold (82°F).

Primary data include core and skin temperatures, arterial blood pressure and LBNP tolerance time. Secondary variables include skin blood flow and heart rate. After completing visit 1 first, all participants will complete visits 2 through 5 in a randomized order and participants are blinded. The order will be counterbalanced between participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 40 years old
* free of known disease and illness
* Speak English
* Systolic blood pressure <140mmHg
* Diastolic blood pressure <90 mmHg

Exclusion Criteria:

* Currently pregnant or breast feeding
* Individuals with diagnosed with cardiac, respiratory, neurological and/or metabolic illness or disease.
* Currently taking prescribed or over the counter medications known to influence the cardiovascular, pulmonary, renal and/or central nervous system.
* Current use of tobacco or nicotine products
* Any physical limitations that impede completion of the tests, such as exercise tests will also be an exclusion criteria.
* Body mass< 80 pounds body weight
* Appendectomy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Arterial blood pressure | Before and during lower body negative pressure (LBNP) procedure
  During simulated blood loss is the reduction in arterial blood pressure greater with progressive skin heating
Tolerance to simulated blood loss | Lower body negative pressure test duration in all trials.
  Tolerance to LBNP will be quantified using the cumulative stress index (CSI) calculated by summing the time at each level of LBNP multiplied by that level (i.e., 20 mmHg * 3 min + 30 mmHg * 3 min + 40 mmHg * 3 min, etc.) until test termination.

SECONDARY OUTCOMES:
Core temperature | Throughout exercise cold exposure and continuously during LBNP
  Measured using rectal probe or intestinal pill and indicative of change in internal body temperature.
Cutaneous Vascular Conductance | Before and during lower body negative pressure (LBNP) procedure
  Skin blood flow measured using laser Doppler flowmetry (AU) will be referenced relative to arterial blood pressure (mmHg) and expressed as cutaneous vascular conductance (CVC; AU/mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: James Pearson, PhD, Principal Investigator — Univeristy of Colorado Colorado Springs
Locations (1):
- University of Colorado Colorado Springs, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results presented in the publication.
Supporting Information: Study Protocol, ICF
Time Frame: Data may be requested up to 36 months following article publication.
Access Criteria: Data will be made available upon reasonable request. Requests should be directed to jpearso5@uccs.edu. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT06279897/Prot_ICF_000.pdf